CLINICAL TRIAL: NCT06606509
Title: The Chinese Clinical Research Plan for the Survey of Treatment and Metabolic Status of Type 1 Diabetes Mellitus (T1DM).
Brief Title: The Survey of Treatment and Metabolic Status of Type 1 Diabetes Mellitus (T1DM).
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20240514-10
Record Dates: First submitted 2024-08-26; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Continuous Glucose Monitoring (CGN); Glucose fluctuations
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- T1DM patients: Patients with Type 1 Diabetes Mellitus (T1DM) will undergo a series of examinations, including physical examinations, surveys, continuous glucose monitoring, and subcutaneous fat ultrasonography.
  Interventions: Device: Continuous Glucose Monitoring System (GX-01S)

INTERVENTIONS:
Device: Continuous Glucose Monitoring System (GX-01S) — Patients with Type 1 Diabetes Mellitus (T1DM) will receive Continuous Glucose Monitoring System (GX-01S) for seven days.

SUMMARY:
This study is a multicenter cross-sectional research project, planning to enroll 1000 patients with Type 1 Diabetes Mellitus (T1DM). By reviewing clinical data, physical examinations, questionnaires, continuous glucose monitoring, and subcutaneous fat ultrasound, we aim to understand the current status of treatment and metabolism in Chinese T1DM patients and analyze the potential factors that may affect their blood sugar control and metabolic indicators. A cost-effectiveness analysis will be conducted on Chinese T1DM patients using continuous glucose monitoring systems to identify the groups that benefit most from these systems.

DETAILED DESCRIPTION:
This study is a multicenter cross-sectional research project, planning to enroll 1000 patients with Type 1 Diabetes Mellitus (T1DM). This study will collect multicenter data on T1DM patients, including sociodemographic information, anthropometric measurements, glycemic indices (glycated hemoglobin, fasting blood glucose, postprandial blood glucose), acute and chronic complications, other important metabolic indicators (blood lipids, vitamin D), insulin treatment methods, blood glucose monitoring status, diabetes education, diet and exercise, social and psychological support, and extra-pancreatic autoimmune diseases. The aims are: 1. To understand the current state of treatment and glycemic metabolism in Chinese T1DM patients and to analyze the potential factors that may affect their glycemic indices. 2. To understand the current status of continuous glucose monitoring (CGM) usage in Chinese T1DM patients and to analyze the impact of CGM on blood glucose control, acute and chronic complications, and quality of life in T1DM patients. 3. Through cost-benefit analysis, to identify potential beneficiary groups for CGM, providing objective evidence for the demand of this technology to healthcare professionals and diabetes patients; to provide effective information for the formulation of medical insurance reimbursement policies for continuous glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate and be able to sign informed consent
* Patients with type 1 diabetes
* At least one of the following three clinical characteristics must be met: The disease presents initially with diabetic ketoacidosis (DKA) or ketonuria; The presence of islet-related autoantibodies, such as islet cell antibodies, tyrosine phosphatase antibodies, or glutamic acid decarboxylase (GAD) antibodies, is detected positively; Both fasting and postprandial C-peptide levels are ≤0.6 ng/mL.

Exclusion Criteria:

* Other types of diabetes.
* Patients who cannot cooperate with the use of continuous glucose monitoring, clinical data collection, and questionnaire completion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study aims to recruit 1,000 patients with Type 1 Diabetes Mellitus (T1DM) from endocrinology departments across various centers between June 2024 and June 2025, both inpatient and outpatient.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-07 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Current status of blood sugar control in Chinese patients with type 1 diabetes | 3 years
  Using continuous glucose monitoring systems to understand the current status of blood sugar control in Chinese patients with type 1 diabetes; analyzing the possible factors that may affect the glycometabolic indicators of Chinese patients with type 1 diabetes.
Understand the current status of the use of continuous glucose monitoring in China for type 1 diabetes | 3 years
  Understand the current status of the use of continuous glucose monitoring in China for type 1 diabetes, and analyze its impact on blood sugar control, acute and chronic complications, and quality of life for patients with type 1 diabetes
Potential beneficiary groups of continuous glucose monitoring | 3 years
  Through cost-effectiveness analysis, identify the potential beneficiary groups of continuous glucose monitoring to provide objective evidence for the demand for this technology by healthcare professionals and diabetes patients; provide effective information for the formulation of medical insurance reimbursement policies for continuous glucose monitoring.

SECONDARY OUTCOMES:
Current treatment status of Chinese patients with type 1 diabetes | 3 years
  Gain a multi-dimensional understanding of the current treatment status of Chinese patients with type 1 diabetes, including aspects such as blood glucose monitoring, education, drug treatment, nutrition, and social support.
Current status of extra-pancreatic autoimmune diseases in Chinese patients with type 1 diabetes | 3 years
  Current status of extra-pancreatic autoimmune diseases in Chinese patients with type 1 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, Doctor, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (101):
- China (101):
  - Anqing Municipal Hospital, Anqing, Anhui
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Hefei First People's Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of USTC,, Hefei, Anhui
  - The second People's Hospital,wuhu, Wuhu, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Shenzhen Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Childrens Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - University-Town Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University second Affiliated Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Quanzhou First Hospital.Fujian, Quanzhou, Fujian
  - Xiamen Fifth Hospital, Xiamen, Fujian
  - Xiamen Hospital of T.C,M., Xiamen, Fujian
  - Zhangshang Hospital Xiamen University, Xiamen, Fujian
  - Gansu Provincial central Hospital, Gansu, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Affiliated Hospital of Youjiang Medical University for Nationalities, Guangxi, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Guangxi, Guangxi
  - The people's Hospital of Guangxi Zhuang Autonomous Region, Guangxi, Guangxi
  - The Second Affiliated Hospital of Guangxi Medical University, Guangxi, Guangxi
  - The First People's Hospital of Qinzhou, Qinzhou, Guangxi
  - Yulin Red Cross Hospital, Yulin, Guangxi
  - Affiliated Hospital of Guangdong Medical University, Guangdong, Guangzhou
  - GuangZhou Eighth People 's Hospital ,GuangZhou Medical University, Guangzhou, Guangzhou
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangzhou
  - The First Affiliated Hospital of Shantou University Medical College, Guangzhou, Guangzhou
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangzhou
  - The Third Hospital of Guangzhou Traditional Chinese Medical University, Guangzhou, Guangzhou
  - People'S Hospital of Anshun City Guizhou Province, Anshun, Guizhou
  - Maternal and Child Health Hospital of Guiyang City, Guiyang, Guizhou
  - Guiqian International General Hospital, Guizhou, Guizhou
  - the First People'S Hospital of Zunyi, Zunyi, Guizhou
  - The First Hospital Of Qinhuangdao, Qinhuangdao, Hebei
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei
  - The Second Hospital Of Hebe Medical University, Shijiazhuang, Hebei
  - Tangshan City Workers Hospital, Tangshan, Hebei
  - The 2nd Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - Heilongjiang Provincial Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The central hospital of nanyang, Nanyang, Henan
  - First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Xinxiang central hospital, Xinxiang, Henan
  - Henan Provincial Peoples Hospital, Zhengzhou, Henan
  - People'S Hospital of Zhengzhou, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhoukou central hospital, Zhoukou, Henan
  - The central hospital of zhumadian, Zhumadian, Henan
  - Jingmen Central Hospital, Jingmen, Hubei
  - Jingzhou central hospital, Jingzhou, Hubei
  - The central hospital of wuhan, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - the First People'S Hospital of Lianyungang, Lianyungang, Jiangsu
  - Jianhua Ma, Nanjing, Jiangsu
  - Jiangsu province hospital of Chinese Medical, Nanjing, Jiangsu
  - Affiliated hospital of nantong university, Nantong, Jiangsu
  - The first affiliated hospital of soochow university, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Gannan, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Province People's Hospital, Jilin, Jilin
  - The First Hospital of Jilin University, Jilin, Jilin
  - The Second Norman Bethune Hospital of Jilin University, Jilin, Jilin
  - The First Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - The People's Hospital Of Liaoning Province, Shenyang, Liaoning
  - Affiliated Hospital of Inner Mongolia University for the Nationalities, Neimeng, Neimenggu
  - Inner Mongolia Medical University Affiliated Hospital, Neimeng, Neimenggu
  - Ningxia Yikedaxuezongyiyuan Xixueguanbing Hospital, Yinchuan, Ningxia
  - The fifth People's Hospital of Qinghai Province, Qinghai, Qinghai
  - Binzhou People's Hospital, Binzhou, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - People's Hospital Of Rizhao, Rizhao, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Shanghai Tenth People'S Hospital, Shanghai, Shanghai Municipality
  - Tong Ren Hospitalshanghaijiaotong Universityschool Ofmedicine, Shanghai, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Weinan Central Hospital, Weinan, Shanxi
  - The first affiliated hospital of xi'an jiaotong university, Xi’an, Shanxi
  - The second affiliated hospital of xi'an jiaotong university, Xi’an, Shanxi
  - The first hospital of yulin, Yulin, Shanxi
  - Chengdu University Affiliated Hospital, Chengdu, Sichuan
  - Piduoqudierrenmingyiyuan, Chengdu, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region, Xinjiang, Xinjiang
  - The First Affiliated Hospital of Shihezi University Medical School, Xinjiang, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang, Xinjiang
  - Urumqi First People's Hospital, Xinjiang, Xinjiang
  - Xinjiang Construction Corps fourth division hospital, Xinjiang, Xinjiang
  - The Fifth Affiliated Hospital of Xinjiang Medical University, Xinxiang, Xinjiang
  - Yunnan First People's Hospital, Yunnan, Yunnan
  - Yunnan University Affiliated Hospital, Yunnan, Yunnan

IPD SHARING:
Plan to Share IPD: No